CLINICAL TRIAL: NCT02279745
Title: An Open-label Extension Study of Ralinepag in Patients With Pulmonary Arterial Hypertension
Brief Title: Long-term Safety and Efficacy of Ralinepag in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD811-007
Record Dates: First submitted 2014-10-25; First posted 2014-10-31 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ralinepag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Ralinepag (Experimental): Ralinepag immediate-release (IR) capsules of 10, 20, 30, 40, and 100 mcg or extended-release (XR) tablets of 50, 250, and 400 mcg for oral administration.
  Interventions: Drug: Ralinepag

INTERVENTIONS:
Drug: Ralinepag — Active
  Other Names: APD811

SUMMARY:
This study was an open-label extension study to determine the long-term safety and tolerability of ralinepag in subjects with World Health Organization (WHO) Group 1 pulmonary arterial hypertension (PAH) who have completed Study APD811-003, or who were assigned to receive placebo and were discontinued due to clinical worsening.

DETAILED DESCRIPTION:
This study was an open-label extension study to determine the long-term safety and tolerability of ralinepag in subjects with WHO Group 1 PAH who completed Study APD811-003. Subjects who completed Study APD811-003 and met eligibility criteria for Study APD811-007 were enrolled. Additionally, placebo-treated subjects who discontinued study drug treatment due to clinical worsening in Study APD811-003 were permitted to enroll in Study APD811-007, upon approval of the medical monitor, provided that all end of study procedures including right heart catheterization (RHC) were performed per the study protocol. The Week 25 Visit in Study APD811-003 served as the Baseline Visit for Study APD811-007.

All subjects enrolled in Study APD811-007 received open-label treatment with ralinepag. The starting dose and titration schedule were individually determined and in accordance with the starting dose and titration schedule optimized from Study APD811-003. Adjustments in the dose and titration schedule were made according to subject tolerability.

After an individual subject completed Study APD811-003 and that subject's database was locked, subject unblinding occurred. Subjects on active treatment (ralinepag) remained on their current dose and had onsite clinical assessments performed every 3 months until the subject was discontinued from the study.

Subjects in the placebo treatment group underwent a dose titration period until a stable, maximum tolerated dose (MTD) was reached (up to 9 weeks), followed by a treatment period after the MTD was determined during which monthly onsite clinic assessments were performed for the first 3 months and then every 3 months until the subject was discontinued from the study or the study was terminated. Dose reductions could be made at any time for safety reasons. Incremental dose increases were also allowed during the Treatment Period at the discretion of the Investigator (as clinically indicated) and according to the stepwise titration scheme.

Subjects were assessed for clinical worsening during each clinic visit. If clinical worsening was confirmed, the Investigator could have opted to either continue treatment with ralinepag at the current dose, increase the dose of ralinepag, interrupt treatment, or discontinue the subject at his/her discretion.

In addition, attempts were made to contact all subjects at the time of Study APD811-007 termination to assess their vital (mortality) status. After the last subject enrolled in Study APD811-007 completed approximately 6 months of the study, a cumulative all-subject data analysis was performed for all subjects who entered the study. Subjects continued to have visits to the clinic every 3 months until the Sponsor discontinued the study. At the time of the Sponsor's decision to discontinue the study, all ongoing subjects completed an End of Study Visit. A 28-day Follow-up Visit was conducted to ensure appropriate subject safety. Subjects who remained on ralinepag were eligible to transition into the Phase 3 open-label extension study (ROR-PH-303) prior to APD811-007 study termination. For those subjects that did not enroll in Study ROR-PH-303, a 28-day Follow-up Visit was conducted to evaluate ongoing subject safety, including survival status.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document.
* Was willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures and was deemed an appropriate candidate for participation in a long-term extension study.
* Female subjects were nonpregnant, nonlactating, surgically sterile or postmenopausal, or agreed to use an accepted method of birth control for at least 3 months prior to the first dose, during, and for at least 30 days after the last dose of study drug.
* Male subjects were either surgically sterile or agreed to use a condom with spermicide when sexually active with a female partner who was not using an acceptable method of birth control during the study and for 30 days after the last dose of study drug.
* Male and female subjects agreed not to participate in a conception process during the study and for 30 days after the last dose of study drug.
* Fulfilled all eligibility criteria for Study APD811-003 and completed the study as planned.

Subjects who were assigned to placebo in Study APD811-003 and experienced clinical worsening in that study could enroll in Study APD811-007 after completing all end of study procedures per protocol, including RHC, for Study APD811-003 and had their data locked.

Exclusion Criteria:

* Subjects who enrolled in Study APD811-003 and were withdrawn from study drug treatment due to any adverse event (AE), serious adverse event (SAE), or subjects who did not complete Study APD811003, with the exception made for placebo-treated subjects who experienced a clinical worsening event.
* Female •subjects who wished to become pregnant.
* Systolic blood pressure <90 mmHg at Baseline.
* Other severe acute or chronic medical or laboratory abnormalities that could have increased the risk associated with study participation or investigational product administration or interfered with the interpretation of study results and, in the judgment of the investigator, would have made the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Cardiac and Vascular Center, Anschutz Inpatient Pavilion, Aurora, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Chest Medicine Associates, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston University Medical Center General Clinical Research Unit (GCRU), Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - UC Health, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - Martha Morehouse Medical Pavilion, Columbus, Ohio
  - UPMC, Presbyterian, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
- Australia (5):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - St Vincent's Hospital, Fitzroy, Victoria
  - Fiona Stanley Hospital, Murdoch
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment "National Heart Hospital" EAD, Clinic of Cardiology, Sofia
  - Multiprofile Hospital for Active Treatment " St. Anna", Sofia AD, Cardiology Clinic, Sofia
- Czechia (2):
  - Department of Internal Medicine I - Cardiology, University Hospital Olomouc, Olomouc
  - Second Internal Clinic - Clinic of Cardiology and Angiology, 1st Faculty of Medicine, Charles University in Prague, General University Hospital in Prague, Prague
- Hungary (5):
  - Gottsegen Gyorgy Orszagos Kardiológiai lntézet - National Institute of Cardiology, Department of Adult Cardiology, Budapest
  - Semmelweis University, Department of Pulmonology - Semmelweis Egyetem Pulmonológiai Klinika, Budapest
  - University of Szeged Faculty of Medicine, 2nd Department of Medicine and Cardiology Center, Albert Szent-Györyi Clinical Center - SZTE ÁOK Szent-Györgyi A lbert Klinikai Központ I I. sz. Belgyógyászati Klini ka és Kard ilógiai Központ, Budapest
  - University of Pecs, Medical School, Heart Institute - Pécsi Tudományegyetem, Klinikai Központ, Szívgyógyászati Klinika, Budapest
  - University of Derecen Clinical Research Center Cardiology and Cardiac Surgery Department - Debreceni Egyetem Klinikai Kozpont Kardiologiai es Szivsebeszeti Klinika, Debrecen
- Poland (3):
  - Medical University of Bialystok Clinical Hospital Cardiology Clinic - Uniwersytecki Szpital Kliniczny, Klinika Kardiologii z Oddziałem Intensywnego Nadzoru Kardiologicznego, Krakow
  - John Paul II Hospital in Cracov Department of Cardiac and Vascular Diseases - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Oddział Kliniczny Chorób Serca i Naczyń, Krakow
  - Biegański Provincial Specialist Hospital Department of Cardiology - Wojewódzki Szpital Specjalistyczny im. dr Wł. Biegańskiego w Lodzi, Oddział Kardiologiczny, Lodz
- Romania (3):
  - "Prof. Dr. C.C. Iliescu" Institute of Cardiovascular Diseases, Department of Clinic Cardiology III - Institutul de Urgenţă pentru Boli Cardiovasculare "Prof. Dr. C.C. Iliescu", Secţia Clinica Cardiologie fIJ, Bucharest
  - "Marius Nasta" Institute of Pneumoftiziology, Department of Pneumoftiziology IV - Institutul de Pneumoftiziologie "Marius Nasta", Sectia Clinica Pneumoftiziologie IV, Bucharest
  - "Dr. Victor Babes" Clinic Hospital for Infesctious Diseases and Pneumoftiziology, Department of Clinic Pneumology II, Timișoara
- Serbia (3):
  - Clinical Centre of Serbia (CCS), Cardiology Clinic - Klinicki Centar SrЬije, Klinika za kardiologiju, Belgrade
  - Кlinicko-bolnicki Centar Zemun, Кlinika za internu medicinu, Sluzba za kardiologiju, Belgrade
  - Institut za plucne bolesti Vojvodine Sremska Kamenica, Klinika za urgcntnu pulmologiju, Odeljcnje intenzivne nege - Institute of Pulmonary Diseases of Vojvodina Sremska Kamenica (IPDVSK), The Clinic for Urgent Pulmonology, ICU - Intensive Care Unit, Kamenitz
- Slovakia (2):
  - Department of Heart Failure and Transplantation, National Institute of Cardiovascular Diseases - Oddelenie zlyhávania a transplantácie srdca, Národný ústav srdcových a cievnych chorôb, a.s., Bratislava
  - Cardiology department, East Slovak Institute for Cardiovascular Diseases - Kardiologické oddelenie Klinika kardiológie , Východoslovenský ústav srdcových a cievnych chorôb, a.s, Košice
- Spain (3):
  - Clinic Hospital of Barcelona, Department of Pneumology, Barcelona
  - General University Hospital Vall d'Hebron, Department of Pneumology, Barcelona
  - Hospital 12th of October, Department of Cardiology, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Ralinepag: Ralinepag immediate-release (IR) capsules of 10, 20, 30, 40, and 100 mcg or extended-release (XR) tablets of 50, 250, and 400 mcg for oral administration were provided. The starting dose and titration schedule were determined for each subject in accordance with the starting dose and titration schedule optimized from Study APD811-003. Subjects in the placebo treatment group in Study APD811-003 underwent a dose titration period (up to 9 weeks) with ralinepag until a stable maximum tolerated dose (MTD) was reached.
  Ralinepag: Active
Period: Overall Study
Arm/Group | Oral Ralinepag
Started | 45
Completed | 25
Not Completed | 20
Not completed — Adverse Event | 7
Not completed — Death | 6
Not completed — Clinical Worsening as Defined by Protocol | 2
Not completed — Withdrawal by Subject | 2
Not completed — Pregnancy | 1
Not completed — Study Non-compliance | 1
Not completed — Did Not Transition to Study ROR-PH-303 | 1

BASELINE CHARACTERISTICS:
Groups:
- Oral Ralinepag: Ralinepag IR capsules of 10, 20, 30, 40, and 100 mcg or XR tablets of 50, 250, and 400 mcg for oral administration were provided. The starting dose and titration schedule were determined for each subject in accordance with the starting dose and titration schedule optimized from Study APD811-003. Subjects in the placebo treatment group in Study APD811-003 underwent a dose titration period (up to 9 weeks) with ralinepag until a stable MTD was reached.
  Ralinepag: Active
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 51.0 [20 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 42
  More than one race | 0
  Unknown or Not Reported | 1
Time Since Pulmonary Arterial Hypertension (PAH) Diagnosis [Median (Full Range); unit: years] | 2.30 [0.8 to 16.0]
Etiology of PAH [Count of Participants; unit: Participants]
  Idiopathic PAH | 23
  Heritable PAH | 4
  Drug or Toxin Induced PAH | 2
  PAH Associated with Other Disease | 16
6-Minute Walk Distance (6MWD) at Baseline [Median (Full Range); unit: meters] | 425.0 [158 to 696]
World Health Organization (WHO) Functional Class at Baseline [Count of Participants; unit: Participants] — I: PH but without limitation of physical activity; physical activity without undue dyspnea or fatigue, chest pain or near syncope.
  II: PH with slight limitation of physical activity; physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  III: PH with marked limitation of physical activity; less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope.
  IV: PH with inability to carry out any physical activity without symptoms. Signs of right heart failure. Dyspnea and/or fatigue at rest. Discomfort is increased by any physical activity.
  Participants
    I | 3
    II | 32
    III | 10
N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) at Baseline [Median (Full Range); unit: pg/mL] | 357.60 [53.4 to 4309.3]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance
Description: Pulmonary vascular resistance was collected by right heart catheterization (RHC).
Time Frame: At 1 or 2 years after the subject enrolled into the study, pending their last RHC prior to Protocol Amendment 2.
Population: The number of subjects varied at post-baseline assessments due to the timing of the assessments relative to the subjects' time on study drug.
Measure: Median (Full Range); unit: dynes.sec/cm5
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 31
dynes.sec/cm5 | -52.2 [-573 to 846]

2. Secondary Outcome: Time From Randomization to the First Protocol-defined Clinical Worsening Event
Description: Clinical worsening events were defined as death, or onset of a treatment-emergent adverse event (AE) with a fatal outcome occurring ≤14 days after treatment discontinuation; hospitalization for worsening PAH, heart-lung or lung transplant, or atrial septostomy; necessity of addition (or dose change) of any prostacyclin/prostacyclin analogue, phosphodiesterase type 5 inhibitor (PDE5-I) or soluble guanylate cyclase (sGC), or endothelin receptor antagonist (ERA); and the combined occurrence of a decrease in 6-Minute Walk Distance (6MWD) by at least 20% from Baseline, confirmed on two 6-Minute Walk Tests (6MWTs) on different days; worsening in WHO/New York Heart Association (NYHA) Functional Class (FC) from Baseline; and appearance of or worsening of signs/symptoms of right heart failure that did not respond to optimized oral diuretic therapy.
Time Frame: From Baseline to 28 days following discontinuation of study drug, up to 235 weeks.
Population: Safety Population
Measure: Median (Full Range); unit: weeks
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 45
weeks | 56.50 [16.9 to 136.6]

3. Secondary Outcome: Change From Baseline in 6MWD
Description: 6MWD was measured at Baseline (prior to starting study drug) and every 3 months thereafter including the End of Study Visit.
Time Frame: From Baseline to discontinuation of study drug, up to 235 weeks
Population: The number of subjects varied from month to month based on total study population at the time of each visit.
Measure: Median (Full Range); unit: meters
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 45
meters
  Month 3: number analyzed (Participants) | 43
  Month 3 | 20.9 [-75 to 115]
  Month 6: number analyzed (Participants) | 42
  Month 6 | 17.6 [-118 to 90]
  Month 9: number analyzed (Participants) | 36
  Month 9 | 22.8 [-88 to 140]
  Month 12: number analyzed (Participants) | 38
  Month 12 | 28.5 [-126 to 138]
  Month 15: number analyzed (Participants) | 34
  Month 15 | 16.2 [-91 to 143]
  Month 18: number analyzed (Participants) | 33
  Month 18 | 16.0 [-100 to 179]
  Month 21: number analyzed (Participants) | 34
  Month 21 | 32.0 [-162 to 175]
  Month 24: number analyzed (Participants) | 33
  Month 24 | 41.0 [-111 to 237]
  Month 27: number analyzed (Participants) | 30
  Month 27 | 38.5 [-141 to 239]
  Month 30: number analyzed (Participants) | 29
  Month 30 | 21.0 [-159 to 267]
  Month 33: number analyzed (Participants) | 24
  Month 33 | 17.0 [-80 to 237]
  Month 36: number analyzed (Participants) | 15
  Month 36 | 47.0 [-60 to 123]
  Month 39: number analyzed (Participants) | 12
  Month 39 | 24.0 [-180 to 105]
  Month 42: number analyzed (Participants) | 11
  Month 42 | 53.0 [-162 to 112]
  Month 45: number analyzed (Participants) | 8
  Month 45 | 20.5 [-160 to 100]
  Month 48: number analyzed (Participants) | 5
  Month 48 | 1.0 [-160 to 57]
  Month 51: number analyzed (Participants) | 1
  Month 51 | -120 [-120 to -120]
  End of Study (Time of Discontinuation of Study by Sponsor): number analyzed (Participants) | 31
  End of Study (Time of Discontinuation of Study by Sponsor) | 37.0 [-327 to 170]

4. Secondary Outcome: Change From Baseline in WHO/NYHA FC
Description: WHO/NYHA FC was measured at Baseline (prior to starting study drug) and every 3 months thereafter including at the End of Study and 28-Day Follow-up Visits. FC recorded as I, II, III, or IV based on the following:
  I: PH but without limitation of physical activity; physical activity without undue dyspnea or fatigue, chest pain or near syncope.
  II: PH with slight limitation of physical activity; physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  III: PH with marked limitation of physical activity; less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope.
  IV: PH with inability to carry out any physical activity without symptoms. Signs of right heart failure. Dyspnea and/or fatigue at rest. Discomfort is increased by any physical activity.
Time Frame: From Baseline to 28 days following discontinuation of study drug, up to 235 weeks
Population: The number of subjects varied from month to month based on total study population at the time of each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 45
Participants
  Month 3: number analyzed (Participants) | 44
  Month 3: Improved | 1
  Month 3: No Change | 43
  Month 3: Deteriorated | 0
  Month 6: number analyzed (Participants) | 42
  Month 6: Improved | 2
  Month 6: No Change | 37
  Month 6: Deteriorated | 3
  Month 9: number analyzed (Participants) | 40
  Month 9: Improved | 1
  Month 9: No Change | 36
  Month 9: Deteriorated | 3
  Month 12: number analyzed (Participants) | 39
  Month 12: Improved | 0
  Month 12: No Change | 37
  Month 12: Deteriorated | 2
  Month 15: number analyzed (Participants) | 36
  Month 15: Improved | 0
  Month 15: No Change | 33
  Month 15: Deteriorated | 3
  Month 18: number analyzed (Participants) | 34
  Month 18: Improved | 2
  Month 18: No Change | 31
  Month 18: Deteriorated | 1
  Month 21: number analyzed (Participants) | 34
  Month 21: Improved | 0
  Month 21: No Change | 30
  Month 21: Deteriorated | 4
  Month 24: number analyzed (Participants) | 33
  Month 24: Improved | 2
  Month 24: No Change | 28
  Month 24: Deteriorated | 3
  Month 27: number analyzed (Participants) | 32
  Month 27: Improved | 2
  Month 27: No Change | 28
  Month 27: Deteriorated | 2
  Month 30: number analyzed (Participants) | 29
  Month 30: Improved | 2
  Month 30: No Change | 23
  Month 30: Deteriorated | 4
  Month 33: number analyzed (Participants) | 25
  Month 33: Improved | 1
  Month 33: No Change | 21
  Month 33: Deteriorated | 3
  Month 36: number analyzed (Participants) | 16
  Month 36: Improved | 1
  Month 36: No Change | 13
  Month 36: Deteriorated | 2
  Month 39: number analyzed (Participants) | 13
  Month 39: Improved | 1
  Month 39: No Change | 11
  Month 39: Deteriorated | 1
  Month 42: number analyzed (Participants) | 11
  Month 42: Improved | 0
  Month 42: No Change | 10
  Month 42: Deteriorated | 1
  Month 45: number analyzed (Participants) | 8
  Month 45: Improved | 1
  Month 45: No Change | 6
  Month 45: Deteriorated | 1
  Month 48: number analyzed (Participants) | 5
  Month 48: Improved | 1
  Month 48: No Change | 4
  Month 48: Deteriorated | 0
  Month 51: number analyzed (Participants) | 2
  Month 51: Improved | 0
  Month 51: No Change | 2
  Month 51: Deteriorated | 0
  End of Study (Time of Discontinuation of Study by Sponsor): number analyzed (Participants) | 35
  End of Study (Time of Discontinuation of Study by Sponsor): Improved | 2
  End of Study (Time of Discontinuation of Study by Sponsor): No Change | 29
  End of Study (Time of Discontinuation of Study by Sponsor): Deteriorated | 4

5. Primary Outcome: Change From Baseline in Cardiac Output
Description: Cardiac output was collected by right heart catheterization (RHC).
Time Frame: At 1 or 2 years after the subject enrolled into the study, pending their last RHC prior to Protocol Amendment 2.
Population: as for outcome 1
Measure: Median (Full Range); unit: L/min
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 31
L/min | -0.0 [-2 to 5]

6. Primary Outcome: Change From Baseline in Cardiac Index
Description: Cardiac index was collected by right heart catheterization (RHC).
Time Frame: At 1 or 2 years after the subject enrolled into the study, pending their last RHC prior to Protocol Amendment 2.
Population: as for outcome 1
Measure: Median (Full Range); unit: L/min/m2
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 31
L/min/m2 | 0.0 [-1 to 3]

7. Primary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure
Description: Mean pulmonary arterial pressure was collected by right heart catheterization (RHC).
Time Frame: At 1 or 2 years after the subject enrolled into the study, pending their last RHC prior to Protocol Amendment 2.
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Oral Ralinepag
Number analyzed (Participants) | 31
mmHg | -2.0 [-23 to 18]

ADVERSE EVENTS:
Time Frame: AEs were recorded for each subject throughout the course of the study from Baseline to 28 days following discontinuation of study drug (up to 235 weeks).
Description: Monitoring of AEs was continued up to 30 days after cessation of study drug administration. If an AE was not resolved or stabilized within 30 days, the Sponsor in consultation with the Investigator decided whether to continue to monitor the AE or close out the event in the database if no further follow-up was necessary. Serious adverse events (SAEs) were monitored until resolution or stabilization.
Groups:
- Oral Ralinepag: Ralinepag IR capsules of 10, 20, 30, 40, and 100 mcg or XR tablets of 50, 250, and 400 mcg for oral administration were provided. The starting dose and titration schedule were determined for each subject in accordance with the starting dose and titration schedule optimized from Study APD811-003. Subjects in the placebo treatment group in Study APD811-003 underwent a dose titration period (up to 9 weeks) with ralinepag until a stable MTD was reached.
  Ralinepag: Active
  There was only 1 active dose group in this open-label study (oral ralinepag). Subjects included in this study received ralinepag and completed previous Study APD811-003, or received placebo and discontinued Study APD811-003 due to clinical worsening. All subjects enrolled in Study APD811-007 received open-label treatment with oral ralinepag IR or XR formulations. The starting dose and titration schedule were individually determined in accordance with the starting dose and titration schedule optimized during Study APD811 003. Adjustments in the dose and titration schedule were made according to subject tolerability.
Arm/Group | Oral Ralinepag
All-Cause Mortality (participants affected / at risk) | 8/45
Serious Adverse Events (participants affected / at risk) | 21/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ralinepag (N=45)
Right ventricular failure (Cardiac disorders) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Ralinepag (N=45)
Anaemia (Blood and lymphatic system disorders) | 8 (12)
Palpitations (Cardiac disorders) | 5 (5)
Right ventricular failure (Cardiac disorders) | 6 (8)
Cardiac failure (Cardiac disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 17 (27)
Nausea (Gastrointestinal disorders) | 14 (25)
Vomiting (Gastrointestinal disorders) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 7 (8)
Oedema peripheral (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 3 (3)
Influenza (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 4 (5)
Bronchitis (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 4 (6)
Urinary tract infection (Infections and infestations) | 4 (7)
Respiratory tract infection (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (6)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 6 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Iron deficiency (Metabolism and nutrition disorders) | 5 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 15 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6)
Headache (Nervous system disorders) | 29 (60)
Dizziness (Nervous system disorders) | 8 (15)
Syncope (Nervous system disorders) | 3 (5)
Presyncope (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Flushing (Vascular disorders) | 12 (16)
Hypotension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT02279745/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT02279745/SAP_001.pdf